CLINICAL TRIAL: NCT02227602
Title: The Mango Consumption Improves Biomarkers for Inflammation in Inflammatory Bowel Disease Patients
Brief Title: Anti-Inflammatory Effects of Mango Polyphenolics in Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Susanne Talcott, PhD, Associate Professor, Nutition & Food Science, Texas A&M University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TexasAMU-IRB2013-0541F
Record Dates: First submitted 2014-06-04; First posted 2014-08-28 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Intestinal Diseases; Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Intestinal Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mango (Experimental): Mango polyphenolics
  Interventions: Drug: Mango polyphenolics

INTERVENTIONS:
Drug: Mango polyphenolics — Frozen mango pack will be provided (200~400g per day).

SUMMARY:
Bioactive compounds from mango are bioavailable and their anti-inflammatory efficacy has been demonstrated in animals and humans. However, the efficacy of mangoes has not previously been compared with respect to mild inflammatory bowel disease. In order to justify future pharmacokinetic and pharmacodynamic analyses in human clinical trials, a pilot assessment to determine efficacy in preventing or resolving Inflammatory bowel disease is a necessary step. Therefore, in this aim we will determine the clinical relevance of mango as an adjuvant treatment to conventional therapy in Inflammatory bowel disease . The effects of mango with common drug treatment in mild-moderate Inflammatory bowel disease will be compared to the drug-treatment alone. If mango or any other polyphenolic-rich food could be identified as helpful in shortening or reducing severity of episodes of inflammatory bowel disease, the addition of polyphenolics to conventional drug treatment in Inflammatory bowel disease would have a significant impact on public health.

DETAILED DESCRIPTION:
Rationale and Significance : Bioactive compounds from mango are bioavailable and their anti-inflammatory efficacy has been demonstrated in animals and humans. However, the efficacy of mangoes has not previously been compared with respect to mild inflammatory bowel disease. In order to justify future pharmacokinetic and pharmacodynamic analyses in human clinical trials, a pilot assessment to determine efficacy in preventing or resolving IBD is a necessary step. Therefore, in this aim we will determine the clinical relevance of mango as an adjuvant treatment to conventional therapy in IBD. The effects of mango with common drug treatment in mild-moderate IBD will be compared to the drug-treatment alone. If mango or any other polyphenolic-rich food could be identified as helpful in shortening or reducing severity of episodes of inflammatory bowel disease, the addition of polyphenolics to conventional drug treatment in IBD would have a significant impact on public health.

The clinical study will be designed in subjects with mild-moderate active Crohn's disease (CD) or mild to moderate ulcerative colitis (UC). This study will be carried out with up to 8 weeks of mango treatment. Subjects with inflammatory bowel disease (IBD; CD or UC) will be performed at the Ertan Digestive Disease Center, Houston, TX, or Texas A&M University, College Station, TX. Patients may be recruited by advertisement (letters, emails, flyers, newspapers) or during standard of clinical care clinics: a) patients coming in for their regular, e.g. semi-annual or annual routine colonoscopy, b) UC or CD-related pain or symptoms, c) individuals presenting with diarrhoea that may be due to Crohn's disease or UC may also be recruited. Informed written consent will be obtained by the research personnel before the study begins. Approximately 90 individuals are expected to enroll in the study in order to obtain 60 subjects completing this study (considering screening failure and potential drop-outs). We expect a maximum of 90 subjects for the initial screening since many of these will be preselected from existing patient files.

This study is designed to incorporate standard of care routine exams as performed within the division of gastroenterology. During the initial screening, the inclusion criteria of patients will be assessed using the clinical indices. it will be performed a screening in which above listed inclusion criteria and hemoglobin, and exclusion parameters and height, weight, calculation of BMI in kg/ (height in meters)2, albumin and C-reactive protein will be assessed due to the high correlation to IBD-activity (>45 mg/L). Subjects will be asked to give a stool sample that has to take place within 1 week before any endoscopic procedure is scheduled and laxatives are taken by the patients in preparation for the procedure.

Study Treatments: Standard of clinical care + 200-400g of Mango b.i.d - t.i.d.,frozen or as smoothie.

This study will be carried out as a pilot study with up to 8 weeks of mango treatment in addition to a list of standard of clinical care drugs. Subjects will be asked to record the exact amount consumed each day. Subjects who skip less than 1 day of mango consumption per week or less than 8 days over the entire period of 8 weeks of mango consumption will not be excluded from this study. Subjects will consume their regular diet but reduce the intake of plant-based dietary supplements which contain secondary plant compounds such as resveratrol, quercetin, tannins, and also reduce their carbohydrate-derived energy by the same amount which is supplied through their mango consumption. Patients that are not receiving the mango will consume their regular diet, which will be controlled for basic nutrients contained in the mango treatment. The mango treatment will start either on this first study day, or as soon as subjects can be classified within the inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 18-79 years (see Protection of Human Subjects)
* Treated with mesalamine or any mesalamine derivate, e.g.Asacol, Apriso, Asacol, Canasa, Lialda, Pentasa, Rowasa orally or rectally as standard of clinical care in the treatment of their symptoms for Inflammatory bowel disease
* Treated using biologic immune-modulators including but not limited to: Infliximab, Adalimumab, Certolizumab, Natalizumab, azathioprine.
* Additionally, patients may be on steroids (prednisone 10mg, budesonide 9mg)
* Subjects must have been on a stable drug-regiment for at least 3 weeks before study begin.

Exclusion Criteria:

* history of acute cardiac event, stroke, or cancer, within the last 6 months,
* recurrent hospitalizations,
* drug treatment of any of the listed conditions within the last 6 months,
* abuse of alcohol or substance within the last 6 months,
* currently smoking more than 1 pack/week,
* seizures,
* liver or renal dysfunction,
* pregnancy or lactation,
* allergy against mangos,
* hepatitis B, C, or HIV,
* regular exercise (>60 minutes, ≥ 5 times/wk), due to association of antioxidant and anti-inflammatory effects and moderate exercise.
* known lactose intolerance, gluten sensitivity, or celiac disease
* Patients that have upcoming Inflammatory bowel disease-related surgery and Inflammatory bowel disease -related intestinal stricture will also be excluded.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2017-05 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Simple Clinical Colitis Activity Index (SCCAI) | 8 weeks
  * A questionnaire used to assess the severity of symptoms in people who suffer from ulcerative colitis
  * The score ranges from 0 to 19, where active disease is a score of 5 or higher
  * compare changes in the score during the study

SECONDARY OUTCOMES:
Short Inflammatory Bowel Disease Questionnaire (SIBDQ) | 8 weeks
  * A health-related quality of life (HRQoL) tool measuring physical, social, and emotional status
  * All scores were reported with a 7-point scale (Score 1-7, 1 = poor HRQOL, 7 = optimum HRQOL).
  * compare changes in the score during the study
Biomarkers for inflammation : hs-CRP, Nf-kB, Il-6, Il-1b in Plasma (pg/ml) | 8 weeks
  - compare changes in the levels during the study

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Talcott, Ph.D, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, Clinical Lab, Nutrition and Food Science Department, College Station, Texas, United States